CLINICAL TRIAL: NCT01288092
Title: A Phase II Study of Orally Administered BEZ235 Monotherapy in Patients With Hormone Receptor Positive, HER2 Negative, Metastatic Breast Cancer, With or Without PI3K Activated Pathway
Brief Title: BEZ235 Trial in Patients With HER2-(Human Epidermal Growth Factor Receptor 2 Negative) /HR+ (Hormonal Receptor Positive) Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235B2201; 2010-024394-39 (EudraCT Number)
Record Dates: First submitted 2011-01-19; First posted 2011-02-02 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; HER2 negative; HR positive; PI3K pathway; no more than 2 prior lines of chemotherapy; Metastatic Breast Cancer(MBC)
MeSH Terms: conditions — Breast Neoplasms | interventions — dactolisib

ARMS (1):
- BEZ235 (Experimental)
  Interventions: Drug: BEZ235

INTERVENTIONS:
Drug: BEZ235

SUMMARY:
This is a prospective, multi-center, open-label, single arm, phase II study with a 2-stage design and Bayesian interim monitoring to investigate the safety and efficacy of BEZ235 in patients with progressive metastatic HR+ HER2- breast cancer who have received at least one prior line of endocrine therapy and two to three prior lines of chemotherapy for metastatic disease. Patients will be stratified into 3 groups according to their PI3K (phosphatidylinositol 3-Kinase) pathway activation status.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years
* ECOG performance status ≤ 2
* Histologically and/or cytologically confirmed diagnosis of breast cancer presenting with metastatic disease (hormone receptor positive and HER2 negative)
* Known PI3K activation status (defined by PIK3CA (Phosphoinositide-3-kinase, catalytic, alpha polypeptide) mutation and PTEN PTEN (Phosphatase and Tensin Homolog) mutation/expression)
* Prior treatment with at least one prior line of endocrine therapy and at least two and no more than three prior lines of chemotherapy for metastatic breast cancer
* Objective and radiologically confirmed progression of disease after prior treatment and at least one measurable lesion as per RECIST
* Adequate bone marrow and organ function

Exclusion Criteria:

* Previous treatment with PI3K and/or mTOR inhibitors
* Symptomatic Central Nervous System (CNS) metastases
* Concurrent malignancy or malignancy in the last 5 years prior to start of study treatment
* Wide field radiotherapy ≤ 28 days or limited field radiation for palliation ≤ 14 days prior to starting study drug
* Active cardiac disease (e.g. Left Ventricular Ejection Fraction (LVEF) < 50%, QTcF > 480 msec on screening ECGelectrocardiogram (ECG), unstable angina pectoris, ventricular, supraventricular or nodal arrhythmias)
* Inadequately controlled hypertension
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BEZ235
* Treatment at start of study treatment with drugs with a known risk to induce Torsades de Pointes, moderate and strong inhibitors or inducers of isoenzyme CYP3A4, warfarin and coumadin analogues, LHRH agonists
* History of photosensitivity reactions to other drugs
* Pregnant or nursing (lactating) woman

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate after 16 weeks of treatment | 16 weeks after the first BEZ235 administration

SECONDARY OUTCOMES:
determine the efficacy of BEZ235 (objective response rate) | about 6 months
evaluate the clinical benefit rate of BEZ235 | about 6 months
evaluate the time to response | about 6 months
evaluate the Progression Free Survival Rate at 16-week & 24-week using the Kaplan-Meier method | 16-week & 24-week after the first BEZ235 administration
evaluate safety of BEZ235 (frequency and severity of Adverse Events, abnormal laboratory values, other safety data as appropriate) | 30-35 days after treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Investigative Site